CLINICAL TRIAL: NCT03481582
Title: Effect of Nitric Oxide Donors on Uterine and Subendometrial Blood Flow in Patients With Unexplained Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rehab Mohamed Abdelrahman, lecturer of obstetric and gynaecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Record Dates: First submitted 2018-03-19; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Polycystic Ovary Syndrome; Infertility, Female
Keywords: Nitroglycerin Trans-dermal Patch
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility, Female | interventions — Nitroglycerin

STUDY DESIGN:
Intervention Model Description: 90 female patients will be divided into 3 equal groups:
  * Group I: 30 female patients with unexplained infertility.
  * Group II: 30 female patients with unexplained infertility will receive nitroglycerin trans-dermal patch.
Who Masked: Participant, Care Provider
Masking Description: * After enrollment, participants would be given the next available number in a computer generated randomization plan .
  * Allocation concealment (among unexplained infertile groups):
  Opaque, serially-numbered, sealed envelopes will enclose the letter corresponding to the group the patient will follow. Envelopes will be opened when the patient is enrolled and she will receive the intervention accordingly.
  -Blinding The study design precludes neither participant nor the doctor will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group without nitroglycerin (Active Comparator): They will be subjected to TV ultrasound for folliculometry till maturation of the follicle ≥18mm then Three dimensional power Doppler will be used to assess the uterine and sub-endometrial blood flow.
  Interventions: Device: Three dimensional power doppler
- Group with nitroglycerin (Experimental): They will receive (nitrodermal®) 5 mg (patch) from 2nd day of cycle till maturation of the follicles ≥ 18 mm then Three dimensional power Doppler will be used to assess the uterine and sub-endometrial blood flow.
  Interventions: Drug: Nitroglycerin; Device: Three dimensional power doppler

INTERVENTIONS:
Drug: Nitroglycerin — (nitrodermal®) 5 mg (patch)as a source of Nitric oxide from 2nd day of cycle till maturation of the follicles ≥ 18 mm just for one cycle.
  Other Names: nitrodermal patch
  Arms: Group with nitroglycerin
Device: Three dimensional power doppler — Once the follicle reached ≥18 mm 3D power Doppler will be used to assess the uterine and subendometrial blood flow

SUMMARY:
The purpose of the study to evaluate effect of nitroglycerin trans-dermal patches on uterine and sub-endometrial blood flow in women with unexplained infertility.

DETAILED DESCRIPTION:
90 female patients will be divided into 2 equal groups:

* Group I: 30 female patients with unexplained infertility.
* Group II: 30 female patients with unexplained infertility will receive nitroglycerin trans-dermal patch.

All subjects will be subjected to the following:

* Proper history taking on past medical history, menstrual history and infertility workup.
* Proper examination (general, abdominal and local examinations)
* Investigations to diagnose unexplained infertility ( male partner's semen analysis as well as documented ovulation and a patent uterine cavity and Fallopian tubes in the female partner).
* Group II (30 patients with unexplained infertility)will receive: (nitrodermal®) 5 mg (patch)as a source of Nitric oxide from 2nd day of cycle till maturation of the follicles ≥ 18 mm just for one cycle
* All women included in each group will be subjected to trans-vaginal ultrasound for folliculometry till maturation of the follicle ≥18mm.
* Once the follicle reached ≥18 mm 3D power Doppler will be used to assess the uterine and sub-endometrial blood flow.
* All women in each group will be subjected to urinary luteinizing hormone (LH) assay. The urinary LH assay will be started on cycle day 11, and repeated daily till detection of the LH surge.
* Six days after detection of the LH surge, 3D power Doppler will be repeated to assess the uterine and sub-endometrial blood flow.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-35 years.6
2. Normal husband's semen analysis (WHO 2010 Criteria):

   * Count ≥15 million
   * Motility ≥ 32% progressive motility
   * Morphology ≥ 4% normal morphology
3. Documented ovulation ( basal body temperature , mid-luteal serum progesterone ≥3 ng / ml and ultrasound monitoring of ovulation).
4. Patent Fallopian tube and excluding uterine anomalies either by hystero-salpingogram (HSG) and/or laparoscopy.
5. Normal hormonal profile (serum progesterone, E2, F.S.H, LH and T.S.H In the 2ND Day of menstrual cycle)

Exclusion Criteria:

1. Male factor of infertility.
2. Patients with uterine pathology as fibroids.
3. Tubal factor of infertility diagnosed by hysterosalpingography (HSG) or laparoscopy.
4. Patients with any contraindications for NO such as chronic liver and renal disease, known cardiac disease and migraine.
5. Diagnosis of PCO based on Rotterdam criteria, two out of three of the following are required to make the diagnosis (Rotterdam, 2004):

   * Oligo- and/or anovulation.
   * Clinical and/or biochemical signs of hyperandrogenism.
   * Polycystic ovaries (by transvaginal ultrasound): the morphology of PCO has been defined as an ovary with 12 or more follicles measuring 2-9 mm in diameter and/or increased ovarian volume (>10 cm3) (Balen et al, 2003).
6. Conditions that mimic PCOS; disorders that cause oligo/anovulation and/or hyperandrogenism, such as:

   * Thyroid disease.
   * Non classic congenital adrenal hyperplasia.
   * Hyperprolactinemia.
   * Androgen-secreting tumors.
7. Women who had any medical comorbidity (e.g. autoimmune disease or diabetes mellitus) and those who have been using medications to induce ovulation or medications known to affect the VEGF concentration (NSAIDs) were not included in the study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Three dimensional power Doppler | from day 10 of menstrual cycle until the follicle reached ≥18 mm
  Once the follicle reached ≥18 mm 3D power Doppler will be used to assess the uterine and sub-endometrial blood flow

SECONDARY OUTCOMES:
Pregnancy rate | 2 weeks after follicle reached ≥18 mm
  serum B-HCG titre if the patient suffered from amenorrhea

CONTACTS AND LOCATIONS:
Locations (1):
- Department of obstetrics and gynaecology, faculty of medicine, Ain shams university, Cairo, Egypt